CLINICAL TRIAL: NCT04129281
Title: Prospective Active Surveillance Versus Surgery in Thyroid Papillary Microcarcinoma
Brief Title: Active Surveillance Versus Surgery in Thyroid Papillary Microcarcinoma
Acronym: MITICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITICA
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Papillary Microcarcinoma of the Thyroid
Keywords: Papillary Microcarcinoma of the Thyroid; Surgery; Outcome; Follow up
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to surgery or active surveillance. Patients who refuse the randomization process will be followed according to the treatment choice according to clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Other): Surgery
  Interventions: Procedure: Surgery
- Active surveillance (No Intervention): Follow up

INTERVENTIONS:
Procedure: Surgery — Surgery acconding to clinical practice
  Arms: Surgery

SUMMARY:
The primary objective of this study is to evaluate the outcome of two treatment approaches (immediate surgery or close follow-up) in patients with papillary thyroid microcarcinoma (mPTc) .

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the outcome of two treatment approaches (immediate surgery or close follow-up) in patients with papillary thyroid microcarcinoma (mPTc) .

A further objective is to identify events associated with high risk of local recurrence and distant metastases.

Patients will be randomized to surgery or active surveillance. Patients who refuse the randomization process will be followed according to the treatment choice according to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >or =18
* Suspicious nodule < or = or 13 mm in the maximum size of thyroid ultrasound (not older than 3 months after the screening visit)
* Cytology consistent with the TIR4 or TIR 5 class
* Sieric TSH in th standard range (with or without levo-tyroxin therapy)
* Normal string motility to fibrolaringoscopy
* Written informed consent

Exclusion Criteria:

* Ultrasound evidence of suspicious lump located on the posterior side of the lobe close to neurogene structures
* Calcitonin increase above normal levels
* Clinical or instrumental evidence of locoregional lymph node metastases (central or laterocervical compartment) or remote
* any Contraindications to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-01-23 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Quality of life in patient who received either surgery or follow up | 36 months
  EORTC QLQ-C30, a quality of life questionnaires, composed by 30 items graded from1 (not at all) to 4 (very much) within 1 year from the diagnosis

SECONDARY OUTCOMES:
Quality of life in patient who received either surgery or follow up | 36 months
  EORTC QLQ-C30, a quality of life questionnaires, composed by 30 items graded from1 (not at all) to 4 (very much) after 1 year from the diagnosis
Compare the two strategies in terms of anxiety/depression | 36 months
  Evaluate the number of patients developing anxiety/depression (Hospital Anxiety and Depression Scale) (HADS scale, Each item on the questionnaire is scored from 0-3 and) in the two groups
Compare the two strategies in terms of adverse events | 36 months
  Evaluate the number of patients developing adverse events (CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Pezzullo, Principal Investigator — IRCCS Study Principal Investigator
Locations (1):
- Istitute Nazionale Tumori - Fondazione G. Pascale, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No